CLINICAL TRIAL: NCT00077922
Title: A Phase II Clinical Trial of Anti-Tac(Fv)-PE38 (LMB-2) Immunotoxin for Treatment of CD25 Positive Chronic Lymphocytic Leukemia
Brief Title: Anti-Tac(Fv)-PE38 (LMB-2) to Treat Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert Kreitman, M.D., Dr. Robert Kreitman, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040121; 04-C-0121; NCT00080821 (obsolete NCT alias)
Record Dates: First submitted 2004-02-12; First posted 2004-02-13 (Estimated); Results first posted 2012-11-15 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Leukemia; Lymphocytic; Chronic
Keywords: LMB-2; Chronic Lymphocytic Leukemia; CLL; Immunotoxin; Oncology; Lymphocytes; Hematological Disease; Monoclonal Antibody; Neutralizing Antibodies
MeSH Terms: conditions — Leukemia; Bronchiolitis Obliterans Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms; Hematologic Diseases | interventions — B3(Fv)-PE38KDEL recombinant immunotoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LMB-2 in chronic lymphocytic leukemia (Experimental): 40 micrograms/kg every other day (QOD) x 3 every 4 weeks in patients with chronic lymphocytic leukemia, the most prevalent form of adult leukemia.
  Interventions: Drug: LMB-2

INTERVENTIONS:
Drug: LMB-2 — 40 micrograms/kg every other day (QOD) x 3 every 4 weeks

SUMMARY:
This study will evaluate the effectiveness of an experimental drug called LMB-2 for treating chronic lymphocytic leukemia (CLL) in patients who have a protein called cluster of differentiation 25 (CD25) on their cancer cells. LMB-2 is a recombinant immunotoxin. It is made up of two parts: a genetically engineered monoclonal antibody that binds to cancer cells with CD25 on their surface, and a toxin produced by bacteria that kills the cancer cells to which it binds. LMB-2 has killed CD 25-containing cells in laboratory experiments and has caused tumors in mice to shrink. Preliminary studies in humans have shown some effectiveness in shrinking tumors in patients with various types of lymph and blood cancers.

Patients 18 years of age and older with CLL who have CD25 receptor proteins on their cancer cells and whose disease has progressed within 2 years of treatment with fludarabine may be eligible for this study. Candidates are screened with a medical history and physical examination, blood and urine tests, electrocardiogram (EKG), echocardiogram, chest x-ray, computed tomography (CT) scans of the chest, abdomen and pelvis, and a bone marrow biopsy.

Participants receive up to six cycles of LMB-2 therapy. Each 28-day cycle consists of 30-minute infusions of LMB-2 on cycle days 1, 3, and 5. The drug is infused through an intravenous (IV) catheter (plastic tube placed in a vein) or a central venous line-an IV tube placed in a large vein in the neck or chest that leads to the heart. Patients are admitted to the National Institutes of Health (NIH) Clinical Center for the first treatment cycle. If the infusion is well tolerated, subsequent cycles may be given on an outpatient basis. In addition to drug therapy, patients undergo the following procedures:

* Blood draws: Blood is drawn before, during, and after each LMB-2 infusion to measure blood levels of the drug, evaluate its effects on the cancer cells, and monitor side effects. Blood tests are also done before and during each cycle to determine how the immune system is interacting with the drug.
* Disease evaluations: Patients undergo a physical examination, blood tests, chest x-ray, and EKG before each treatment cycle and at follow-up visits. With the patient's permission, CT scans, echocardiogram, and bone marrow biopsies may be repeated before some treatment cycles if these tests prove useful in evaluating the disease response to LMB-2.

Patients may receive up to six cycles of LMB-2 as long as their cancer does not worsen and they do not develop serious side effects. At the end of the treatment cycles, patients will have blood tests done weekly by their local physician, and the results will be sent to the NCI study investigators.

DETAILED DESCRIPTION:
Background:

It is estimated that 30-50% of patients with CLL have tumors that express cluster of differentiation 25 (CD25) (Tac or IL2R). Normal resting T-cells are not sensitive to LMB-2 due to insufficient CD25 expression. LMB-2 is an anti-CD25 recombinant immunotoxin containing variable domains of MAb anti-Tac and truncated Pseudomonas exotoxin. A phase I trial at National Cancer Institute (NCI) found that the maximum tolerated dose (MTD) of LMB-2 was 40 microg/Kg IV given every other day for 3 doses (every other day (QOD) x3) with prophylactic IV fluid. The most common adverse events were transient fever, hypoalbuminemia and transaminase elevations. In that trial, one of eight patients with chronic lymphocytic leukemia had a partial remission. The other seven CLL patients had stable disease. In addition, four of four patients with hairy cell leukemia had responses (1 complete response (CR), 3 partial response (PRs)) and 3 other patients had PRs (1 cutaneous T-cell lymphoma (CTCL), 1 healthy donor (HD), 1 acute T-cell leukemia/lymphoma (ATL)). Because LMB-2 is cytotoxic to cells expressing CD25, CD25+ CLL patients are good candidates for further testing with LMB-2.

Objectives:

The purpose of this study is to determine the activity of anti-Tac(Fv)-PE38 (LMB- 2) in patients with Tac-expressing Chronic Lymphocytic Leukemia (CLL). The primary endpoint of this trial is response rate. We will also evaluate response duration, LMB-2 immunogenicity, pharmacokinetics, toxicity, and monitor soluble Tac levels in the serum.

Eligibility:

CD25 positive CLL or prolymphocytic leukemia (PLL) confirmed by flow cytometry of blood, with either lymphadenopathy, splenomegaly, hepatomegaly, hemoglobin less than 11 g/dl,

or platelets less than 100,000/ul.

Patients must have progression following purine analog or alkylating agent.

Labs required: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 2.5- time upper limit,

albumin greater than or equal to 3, bilirubin less than equal to 2.2 (unless unconjugated greater than or equal to 80%)

and creatinine less than or equal to 1.4 (unless creatinine clearance greater than or equal to 50 ml/min).

Design:

Patients receive LMB-2 40 ug/Kg QOD x3 every 4 weeks in absence of neutralizing antibodies or progressive disease. 1st stage is 16 patients, to expand to 25 if greater than 1 of 16 patients respond.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have histopathological evidence of CD25+ CLL or prolymphocytic leukemia (PLL) confirmed by the NIH pathology department. This requires that at least 50% of the peripheral malignant lymphocytes be CD25 positive by fluorescence activated cell sorting (FACS) with anti-CD25 antibody. Positive expression in a FACS assay is defined as more than 2 times the mean fluorescence intensity (MFI) of the control antibody by FACS, or greater than 400 CD25 sites/cell by FACS or radiolabeled binding assay.

In the three stage modified Rai system, patients must be intermediate or high risk. This means they must have circulating CLL cells and at least one of the following: lymphadenopathy, splenomegaly, hepatomegaly, anemia (Hgb less than 11g/dL), or thrombocytopenia (Plt less than 100,000/ul).

Patients must have had progressive disease after prior standard therapy containing either a purine analog or an alkylating agent.

Patients must not have received systemic cytotoxic chemotherapy within 4 weeks of enrollment or systemic steroids (except stable doses of Prednisone less than or equal to 20 mg/day) within 4 weeks of enrollment.

Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2.

At least 18 years old.

Patients must be able to understand and give informed consent.

Female patients of childbearing potential must have a negative pregnancy test and all patients must use effective contraception (a barrier form of contraception).

The transaminases alanine aminotransferase (ALT) and aspartate aminotransferase (AST) must each be less than or equal to 2.5-times the upper limits of normal. Albumin must be greater than or equal to 3.0 gm/dL. Total bilirubin must be less than or equal to 2.2 mg/dL except in patients with Gilbert's syndrome (as defined by greater than 80% unconjugated bilirubin) it must be less than 5 mg/dl.

The creatinine must be less than or equal to 1.4 mg/dL or the creatinine clearance must be greater than or equal to 50 ml/min as measured from a 24-hour urine collection.

Patients should not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

EXCLUSION CRITERIA:

Patients whose serum neutralizes LMB-2 in tissue culture, due either to anti-toxin or anti-mouse-lgG antibodies. No patient whose serum neutralizes greater than 75% of the activity of 1 micro g/mL of LMB-2 will be treated.

Patients who received LMB-2 on another trial.

Monoclonal antibody therapy within 12 weeks of enrollment.

Patients who are pregnant or breast-feeding.

Patients who are human immunodeficiency virus (HIV) positive.

Patients who have hepatitis C or chronic liver disease. Patients would not be excluded for hepatitis B surface antigen positivity if on Lamivudine.

Patients receiving warfarin for anticoagulation.

Patients with a left ventricular ejection fraction of less than the institutional lower limit of normal.

Patients with a carbon monoxide diffusing capacity (DLCO) less than 55% of normal or an forced expiratory volume 1 (FEV1) less than 60% of normal.

Patients who have active cancer requiring treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-02-29 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2011-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Kreitman, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheson BD, Bennett JM, Grever M, Kay N, Keating MJ, O'Brien S, Rai KR. National Cancer Institute-sponsored Working Group guidelines for chronic lymphocytic leukemia: revised guidelines for diagnosis and treatment. Blood. 1996 Jun 15;87(12):4990-7. No abstract available. PMID 8652811
- [Background] Harris NL, Jaffe ES, Diebold J, Flandrin G, Muller-Hermelink HK, Vardiman J, Lister TA, Bloomfield CD. World Health Organization classification of neoplastic diseases of the hematopoietic and lymphoid tissues: report of the Clinical Advisory Committee meeting-Airlie House, Virginia, November 1997. J Clin Oncol. 1999 Dec;17(12):3835-49. doi: 10.1200/JCO.1999.17.12.3835. PMID 10577857
- [Background] Rai KR, Sawitsky A. A review of the prognostic role of cytogenetic, phenotypic, morphologic, and immune function characteristics in chronic lymphocytic leukemia. Blood Cells. 1987;12(2):327-38. PMID 3304471

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LMB-2 in Chronic Lymphocytic Leukemia
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LMB-2 in Chronic Lymphocytic Leukemia
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.36 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response is measured by the 1996 National Cancer Institute (NCI) Working Group Criteria (NCIWG). Complete response is defined as no hepatomegaly, splenomegaly, or lymphadenopathy by physical examination and appropriate radiographic techniques. Lymph nodes must resolve to <1.0cm of 1-1.5cm at baseline, or <1.5cm if >1.5cm at baseline. Partial response is >=50% decrease in peripheral blood lymphocytes count from the pretreatment baseline value. Progressive disease is >=50% increase in the sum of the products of the greatest perpendicular dimensions of a t least 2 lymph nodes on two consecutive examinations 2 weeks apart (at least 1 node must be >=2cm) or appearance of new palpable lymph nodes. Stable disease is characterized by not meeting the above criteria. For additional details about the NCIWG, see the protocol link module.
Time Frame: Patients were followed for at least 30 days after last treatment. Because the study allows 6 treatment cycles, this can be up to 7 months.
Measure: Number; unit: Participants
Arm/Group | LMB-2 in Chronic Lymphocytic Leukemia
Number analyzed (Participants) | 15
Participants
  Complete Response | 0
  Partial Response | 1
  Progressive Disease | 3
  Stable Disease | 11

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 54 months
Measure: Number; unit: Participants
Arm/Group | LMB-2 in Chronic Lymphocytic Leukemia
Number analyzed (Participants) | 15
Participants | 15

ADVERSE EVENTS:
Time Frame: 54 months
Arm/Group | LMB-2 in Chronic Lymphocytic Leukemia
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 7/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LMB-2 in Chronic Lymphocytic Leukemia (N=15)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Cardiac-ischemia/infarction (Cardiac disorders) | 1 (1)
Cardiac troponin I (cTnI) (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Lung (pneumonia)
Infection (documented clinically or microbiologically) (Infections and infestations) | 2 (2) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Skin (cellulitis)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 1 (1)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Ocular/Visual-Other (Specify, blindness r/t CVA) (Eye disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Obstruction, GU: Ureter (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LMB-2 in Chronic Lymphocytic Leukemia (N=15)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2 (2)
haptoglobin (Blood and lymphatic system disorders) | 2 (5)
Hemoglobin (Blood and lymphatic system disorders) | 9 (71)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (4)
Neutrophils/granulocytes (ANC/AG) (Blood and lymphatic system disorders) | 8 (30)
Platelets (Blood and lymphatic system disorders) | 7 (48)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 3 (3)
Hypotension (Cardiac disorders) | 3 (4)
Pericardial effusion (non-malignant) (Cardiac disorders) | 3 (3)
fibrinogen (Blood and lymphatic system disorders) | 1 (1)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 7 (13)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 11 (23)
Insomnia (General disorders) | 3 (3)
Rigors/chills (General disorders) | 3 (4)
Sweating (diaphoresis) (General disorders) | 2 (2)
Weight gain (General disorders) | 9 (15)
Weight loss (General disorders) | 1 (1)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 5 (5)
Dermatology/Skin - Other (Specify) (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 2 (2)
Heartburn/dyspepsia (Gastrointestinal disorders) | 2 (2)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (12)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 4 (6)
Hemorrhage, GI::Oral cavity (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GU: Bladder (Renal and urinary disorders) | 1 (1)
Hemorrhage, GU: Urinary NOS (Renal and urinary disorders) | 6 (8)
Hemorrhage, pulmonary/upper respiratory: Lung (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory: Nose (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 2 (2)
Febrile neutropenia (Infections and infestations) | 1 (1) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (1) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Catheter-related
Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (1) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L):: Lung (pneumonia)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lip/perioral (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Oral cavity-gums (gingivitis) (Infections and infestations) | 3 (7)
Infection with normal ANC or Grade 1 or 2 neutrophils::Sinus (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 2 (2)
Edema: limb (Blood and lymphatic system disorders) | 10 (19)
Edema::head and neck (Blood and lymphatic system disorders) | 6 (14)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 4 (10)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 11 (49)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 14 (72)
Alkaline phosphatase (Metabolism and nutrition disorders) | 6 (19)
Amylase (Metabolism and nutrition disorders) | 3 (4)
Bicarbonate, serum low (Metabolism and nutrition disorders) | 2 (4)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 5 (13)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 3 (7)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 3 (11)
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 2 (4)
Creatinine (Metabolism and nutrition disorders) | 4 (8)
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 3 (5)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 7 (12)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 3 (8)
Hemoglobinuria (Metabolism and nutrition disorders) | 3 (3)
Lipase (Metabolism and nutrition disorders) | 2 (2)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 6/8 (12)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 8 (26)
Phosphate, serum-high (hyperphosphatemia) (Metabolism and nutrition disorders) | 7 (17)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 4 (9)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 5 (22)
Proteinuria (Metabolism and nutrition disorders) | 3 (3)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 5 (6)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 7 (25)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 3 (4)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 3 (3)
Confusion (Nervous system disorders) | 1 (2)
Dizziness (Nervous system disorders) | 6 (9)
Mood alteration::Anxiety (Nervous system disorders) | 1 (1)
Mood alteration::Depression (Nervous system disorders) | 1 (1)
Neurology-Other (Specify, dizziness) (Nervous system disorders) | 1 (1)
Neuropathy:sensory (Nervous system disorders) | 1 (1)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 2 (2)
Ocular surface disease (Eye disorders) | 2 (2)
Vision-blurred vision (Eye disorders) | 1 (1)
Pain - Other (Specify, extremity, limb) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain: Abdomen NOS (Gastrointestinal disorders) | 1 (1)
Pain: Back (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Chest wall (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pain::Dental/teeth/peridontal (Gastrointestinal disorders) | 1 (1)
Pain: Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Eye (Eye disorders) | 1 (1)
Pain::Head/headache (Nervous system disorders) | 7 (11)
Pain::Middle ear (Ear and labyrinth disorders) | 1 (1)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 6 (9)
Pain::Neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Neuralgia/peripheral nerve (Nervous system disorders) | 2 (2)
Pain::Oral cavity (Gastrointestinal disorders) | 2 (2)
Pain::Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Bladder spasms (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (2)
Flu-like symptoms (General disorders) | 2 (2)
Acute vascular leak syndrome (Vascular disorders) | 7 (12)
Phlebitis (including superficial thrombosis) (Vascular disorders) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2011-07-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT00077922/Prot_SAP_ICF_000.pdf